CLINICAL TRIAL: NCT00135681
Title: Immune Dysregulation in Children and Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 244; P50HL056384 (NIH)
Record Dates: First submitted 2005-08-23; First posted 2005-08-26 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

INTERVENTIONS:
Drug: nedocromil budesonide

SUMMARY:
To immunize both normal and asthmatic subjects with a neoantigen, keyhole limpet hemocyanin (KLH) and observe the type of antibody and T cell response that develops.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a result of a dysregulated immune response to inhaled antigens. The development of an immune response dominated by T cells (Th2) that secrete interleukin 4 (IL-4) and IL-5 results in the constellation of findings associated with asthma, including elevated IgE and increased blood eosinophilia. Epidemiological studies indicate that there are several predisposing factors that may dictate whether asthma may develop in certain individuals including genetic, environmental, and age-related factors. Any one factor alone may not determine whether an inappropriate immune response develops with subsequent development of asthma; rather, asthma likely results from a combination of factors. However, once a Th2 response in the lung has occurred, the hypothesis is that it dominates and results in the development of Th2 response to inhaled neoantigens. Further, the acquired predisposition to a Th2 response may override other preexisting predisposing factors and therefore becomes the prime target for asthma therapy.

DESIGN NARRATIVE:

The study was a subproject in a Specialized Center of Research (SCOR) in Fibrotic Lung Disease from 1997 through 2001. Both normal and asthmatic subjects were immunized with a neoantigen, keyhole limpet hemocyanin (KLH), via intrapulmonary and subcutaneous routes and observed for the type of antibody and T cell response that developed. Furthermore, the effect of inhaled anti-inflammatory medications on primary immune responses to KLH was assessed. Additional studies examined the effect of regional pulmonary Th2 responses on peripheral blood asthma-associated effector cells, basophils and eosinophils. Finally, the investigators determined whether chronic therapy of asthmatic children with either nedocromil or budesonide modulated their immune response to a systemically administered neoantigen, hepatitis B vaccine. These studies were designed to provide important information on the regulation of immune responses in humans with asthma. Furthermore, they helped to determine whether anti-inflammatory medications could inhibit development of a Th2 responses or only prevent inflammatory events downstream from Th2 development.

The subproject had three specific aims. The first was to test the hypothesis that the lower respiratory tracts of asthmatics would respond differently to a neo-antigen. In part A of specific aim 1, the lower respiratory tracts of asthmatics were challenged with KLH. Bronchoalveolar lavage (BAL) was repeated after 12 days and blood samples collected after a number of time points. Immunoglobulins were measured in blood and BAL, and lymphocytes were collected from the BAL and assayed for response to antigen in an in vitro test. In part B, individuals were treated with six weeks of anti-inflammatory therapy after which responses to intrapulmonary antigen were assessed.

Specific aim 2 assessed the role of acute challenge of the lung with antigen on eosinophil and basophil responsiveness. The lung was challenged by intrapulmonary installation of antigen through the bronchoscope and samples were collected from the peripheral blood at various time points. An allergen challenge was performed after six weeks of therapy with nedocromil budesonide or placebo.

In specific aim 3, asthmatic children were tested in two stages. In stage one, a preliminary study was performed in children with relatively mild asthma who were immunized with hepatitis vaccine. Samples were collected at various time points and assayed for antigen-specific antibody. The hypothesis that asthmatic children would have a Th2 type response rather than the Th1 type response in normal children was evaluated by determining times at which samples could be collected from the larger Childhood Asthma Management Program (CAMP) study.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-12; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schuyler (Subproject PI) — University of New Mexico